CLINICAL TRIAL: NCT06538337
Title: Hypofractionated External Beam Radiotherapy With Adaptive Planning for Endometrial and Cervical Cancers (HERA Trial)
Brief Title: Hypofractionated External Beam Radiotherapy With Adaptive Planning for Endometrial and Cervical Cancers
Acronym: HERA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-001976
Record Dates: First submitted 2024-07-22; First posted 2024-08-05 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Endometrial Cancer; Cervical Cancer
Keywords: endometrial; cervical; SBRT
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm, non-randomized, trial of adjuvant SBRT to the pelvis with adaptive planning using CT or MRI guidance for endometrial and cervical cancers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hypofractionated External beam Radiotherapy (Experimental): 5 daily treatment sessions of MRI or CT-Guided Stereotactic Body Radiation Therapy (SBRT).
  Interventions: Radiation: External beam Radiotherapy

INTERVENTIONS:
Radiation: External beam Radiotherapy — Five fractions of radiation therapy using adaptive planning and CT or MRI guidance (6 Gy per fraction) delivered once every other day excluding weekends and holidays
  Other Names: Hypofractionated External beam Radiotherapy

SUMMARY:
After surgery to remove the main endometrial and/or cervical tumor, most women receive radiation therapy. This study uses hypo-fractionated radiation therapy, which is a type of radiation therapy in which the total prescribed dose of radiation is delivered in fewer but larger doses than conventional or standard radiotherapy.

This research study aims to determine if hypo-fractionated radiation therapy given after surgery can improve treatment tolerability (i.e., fewer treatments) with comparable side effects.

Participants will be in the study for about 5 years:

Radiation therapy:

* 5 daily treatment sessions of MRI or CT-Guided Stereotactic Body Radiation Therapy (SBRT).
* Each treatment session will occur on a weekday (typically consecutive weekdays) and will last approximately an hour.

Treatment Follow-Up:

* Check-up Appointment and answer questions at 3 months post RT
* Check-up Appointments with physical exam every 6 months (+/- 4 weeks) for up to 5 years.

DETAILED DESCRIPTION:
The investigators hypothesize that adaptive planning with either computed tomography (CT) or magnetic resonance imaging (MRI) guidance may offer improved SBRT plans for postoperative gynecological cancer patients due to issues with anatomic variation between and during fractions of radiation therapy. Treatment on an MRI-guided linear accelerator with adaptive planning capabilities has been shown to significantly improve acute toxicity in the setting of prostate SBRT compared to conventional linear accelerators.10 The investigators, therefore, propose using adaptive planning with CT- or MRI-guidance to deliver 30 Gy in 5 fraction adjuvant SBRT to the pelvis for endometrial and cervical cancer patients.

Stereotactic Body Radiation Therapy (SBRT) with adaptive planning will be delivered following surgical resection of the primary tumor. Patients will receive 6.0 Gy x 5 fractions delivered once every other day. Patients will not be treated on weekends or holidays as is standard practice for radiation treatments.

Patients will be seen by the radiation oncologist within the first 3 months after completion of radiation therapy. For patients who live a distance far enough away from the University of California at Los Angeles (UCLA) where travel would be challenging for the patient, a phone or telemedicine follow-up will be considered acceptable. After this, follow-up will be performed every 6 months (+/- 4 weeks) for 5 years following completion of radiotherapy. Patients will be followed clinically and/or radiographically per physician discretion.

SCHEMA

Diagnosis of endometrial or cervical cancer

Surgical resection of primary tumor

Multidisciplinary discussion and recommendation for adjuvant radiotherapy to the pelvis

Patient enrollment in HERA clinical trial

Simulation scans to plan post-operative radiotherapy

Five fractions of radiation therapy using adaptive planning and CT or MRI guidance (6 Gy per fraction) delivered once every other day excluding weekends and holidays

Follow-up within 3 months of completion of radiotherapy

Follow-up every 6 months (+/- 4 weeks) until 5 years of completion of radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed endometrial or cervical cancer
* Surgical resection of the primary tumor
* International Federation of Gynecology and Obstetrics (FIGO) Stage IA-IVB endometrial cancer OR FIGO Stage IA-IIA cervical cancer that meets indications for receiving adjuvant pelvic radiotherapy alone as standard of care
* Age ≥ 18 years old
* Karnofsky performance status (KPS) ≥ 60 or Eastern Cooperative Oncology Group (ECOG) 0-2

Exclusion Criteria:

* Must not meet indications for receiving concurrent chemotherapy as standard of care
* Active treatment of a separate malignancy
* History of prior irradiation to the area to be treated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study considers endometrial and cervical cancer which are defined as physically occurring in the uterus and the cervix.
Enrollment: 60 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2031-07-26 (Estimated); Study Completion 2032-07-26 (Estimated)

PRIMARY OUTCOMES:
Evaluate acute radiation toxicity | treatment to 12 weeks after completion of radiotherapy
  Evaluate acute radiation toxicity according to Common Terminology Criteria for Adverse Events, Version 5.0 (CTCAE v5.0). Acute toxicity is defined as treatment-related adverse events occurring within 12 weeks of completion of radiotherapy.

SECONDARY OUTCOMES:
Evaluate patient-reported quality-of-life European Organization for Research and Treatment of Cancer Quality of Life (EORTC QLQ-C30) | treatment to 24 weeks after completion of radiotherapy
  Evaluate patient-reported quality-of-life scores using European Organization for Research and Treatment of Cancer Quality of Life Questionnaires (QLQ) C30 (EORTC QLQ-C30). The EORTC QLQ-C30 is a 30-item instrument designed to assess various aspects of the overall quality of life in patients with cancer. We will collect data pre-treatment and 3, 6-, 12-, 18-, and 24-months post-treatment.
  The EORTC QLQ-C30 uses a 4-point response scale for most items: 1 = not at all, 2 = a little, 3 = quite a bit, and 4 = very much.
  A higher score indicates worse quality of life.
Evaluate patient-reported quality-of-life European Organization for Research and Treatment of Cancer Quality of Life (EORTC QLQ-EN24) | treatment to 24 weeks after completion of radiotherapy
  Evaluate patient-reported quality-of-life scores using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Endometrial Cancer Module (EORTC QLQ-EN24). The EORTC QLQ-EN24 is a 24-item instrument designed to assess various aspects of treatment-related quality of life specifically in patients undergoing treatment for endometrial cancer. We will collect data pre-treatment and 3, 6-, 12-, 18-, and 24-months post-treatment.
  The EORTC QLQ-EN24 uses a 4-point response scale for most items: 1 = not at all, 2 = a little, 3 = quite a bit, and 4 = very much.
  A higher score indicates worse quality of life.
Evaluate late toxicity | 12 weeks after completion of radiotherapy until 5 years after completion of radiotherapy
  Evaluate late toxicity according to Common Terminology Criteria for Adverse Events, Version 5.0 (CTCAE v5.0). Late toxicity is defined as treatment-related adverse events occurring more than 12 weeks after completion of radiotherapy.
Evaluate local control | treatment to 5 years after completion of radiotherapy
  Evaluating control of the treated tumor. Local control will be estimated using Kaplan-Meier analysis at 5 years.
Evaluate regional control | treatment to 5 years after completion of radiotherapy
  Evaluating control of disease within the abdomen and pelvis. Regional control will be estimated using Kaplan-Meier analysis at 5 years.
Evaluate distant metastasis | treatment to 5 years after completion of radiotherapy
  Evaluating the spread of the disease to distant sites. Distant metastasis will be estimated using Kaplan-Meier analysis at 5 years.
Evaluate progression-free survival | treatment to 5 years after completion of radiotherapy
  Evaluating patient survival free from any disease progression (local, regional, or distant). Progression-free survival will be estimated using Kaplan-Meier analysis at 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Puja S. Venkat, MD, Principal Investigator — University of California at Los Angeles
Locations (1):
- University of California at Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided